CLINICAL TRIAL: NCT05587127
Title: A Randomized Controlled Trial of Exposure-Based Cognitive Behavioral Treatment for Avoidant/Restrictive Food Intake in Functional Dyspepsia
Brief Title: Exposure-Based CBT for Avoidant/Restrictive Food Intake in Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Helen B. Murray, PHD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022P001765; K23DK131334-01 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Avoidant/Restrictive Food Intake Disorder; Dyspepsia; Feeding and Eating Disorders; Cognitive Behavioral Therapy; Appetite Regulation; Functional Dyspepsia; Post-prandial Distress Syndrome; Behavioral Medicine
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Dyspepsia; Feeding and Eating Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Subjects will receive cognitive behavioral therapy for functional dyspepsia with avoidant restrictive food intake disorder.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Usual Care (No Intervention): In the usual care condition, participants will be allowed to continue with treatment they are already receiving at the time of randomization, and we will collect detailed data on the nature of these interventions. Participants will be allowed to pursue non study treatments in this condition.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Eight 1-hour sessions delivered weekly via the MGH-approved secure video platform Enterprise Zoom. Skills include: education about gut-brain regulation and weight loss, and regularizing eating to improve hunger and satiety cues; techniques to facilitate weight gain with targets of increased food volume and variety; and plan for maintenance of treatment gains.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Randomized controlled trial of an exposure-based behavioral treatment (CBT) in adults with functional dyspepsia who meet criteria for avoidant/restrictive food intake disorder (ARFID) with weight loss.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized controlled trial (RCT) of a cognitive-behavioral treatment (CBT) compared to usual care as the control with adults with functional dyspepsia who also meet criteria for avoidant/restrictive food intake disorder (ARFID). Participants randomized into the CBT group will receive eight 1-hour sessions delivered weekly via the MGH-approved secure video platform Enterprise Zoom while the usual care group will be allowed to continue with treatment they are already receiving at the time of randomization. Participants in the usual care group will be offered CBT after study participation. We will determine the feasibility and acceptability of the CBT and explore changes in clinical outcomes and preliminary mechanisms.

ELIGIBILITY:
Inclusion Criteria

* Age at least 18 years at screening visit
* Rome IV Functional Dyspepsia post-prandial distress type (with or without epigastric pain syndrome)
* Negative upper endoscopy or upper radiographic GI series to rule out structural/organic cause for FD
* Avoidant/Restrictive Food Intake Disorder (ARFID) diagnosis (by the Structured Clinical Interview for DSM-5; SCID-5 at Screening visit)
* ≥5% weight loss from weight after functional dyspepsia symptom onset (at Screening visit)
* Stable for outpatient care (based on the American Psychiatric Association Practice Guideline for the Treatment of Patients with Eating Disorders)
* No previous history of CBT for functional dyspepsia or ARFID
* Computer/internet webcam access
* Fluency in English
* Stable dose for 30 days if on any medication

Exclusion Criteria

* Inability to provide informed consent
* Presence of other conditions that could explain the patient's symptoms by chart:

Pyloric or intestinal obstruction (by EGD, UGI, or Abdominal CT) Active H.pylori infection (by CLO test or stool antigen test) Active inflammatory bowel disease Eosinophilic gastroenteritis or eosinophilic esophagitis Acute renal failure Chronic renal failure (serum creatinine >3 mg/dL) and/or on hemodialysis or peritoneal dialysis Acute liver failure Any acute gastrointestinal process Any plausible structural or metabolic causes Heartburn as predominant symptom History of peptic ulcer

* Symptom resolution with antisecretory therapy (PPI use for other reasons that did not resolve FD symptoms will be allowed)
* History of gastrointestinal tract surgery (including gastrectomy, gastric bypass surgery, and small or large bowel resection)
* History of any serious medical condition (e.g., cancer)
* Use of narcotic analgesics greater than three days per week
* Current pregnancy or breastfeeding within the last 8 weeks
* Uncontrolled diabetes (indicated by HbA1c ≥7%) by chart
* Intellectual disability by history
* Current substance/alcohol use disorder within the past month
* Current/history of psychosis (by Mini-International Neuropsychiatric Interview (MINI-Screen)
* Current mania (by Mini-International Neuropsychiatric Interview (MINI-Screen) (defined as any manic episodes within the past 12 months)
* Active suicidal ideation (by MINI-Screen)
* Psychiatric disorder that would warrant independent attention (by Mini-International - Neuropsychiatric Interview (MINI-Screen))
* Current enteral or parenteral feeding
* Plans to initiate another psychotherapy or pregnancy in the concurrent study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Enrollment | Throughout study completion, an average of 3 years
  At the end of the study, we will calculate the percentage of participants who consent to initiate the study from the total who are offered.
Assessment completion | Throughout study completion, an average of 3 years
  At the end of the study, we will calculate the percentage of participants who complete all assessments in each CBT and usual care groups.
Retention | Throughout study completion, an average of 3 years
  At the end of the study, we will calculate the percentage of participants who complete at least 6 of the 8 CBT sessions.
Interventionist Fidelity ratings | Throughout study completion, an average of 3 years
  At the end of the study, we will calculate fidelity, which measures the percentage of sessions that 100% of the CBT content was delivered.
Client Satisfaction | Week 12
  The Client Satisfaction Questionnaire (CSQ) is an 8 item self-report measure that assesses treatment satisfaction. Higher scores indicate greater treatment satisfaction.

SECONDARY OUTCOMES:
Short Form Nepean Dyspepsia Inventory (SF-NDI) | Weeks 0, 6, and 12
  The Short Form Nepean Dyspepsia Inventory (SF-NDI) includes a 15 item symptoms checklist to assess functional dyspepsia symptom severity. It also includes 10 items scored on a 5-point Likert scale measuring functional dyspepsia-related quality of life; subscales include interference with daily activities, knowledge/control, tension, work/study, and eating/drinking.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Burton Murray, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States